CLINICAL TRIAL: NCT02436538
Title: Correlation Between Serum Anti-Müllerian Hormone (AMH) Levels & Müllerian Ducts Anomalies in Patients Undergoingintracytoplasmic Sperm Injection (ICSI)
Brief Title: Correlation Between Serum Anti-Müllerian Hormone & Müllerian Ducts Anomalies in Infertility
Status: Completed | Type: Observational
Sponsor: Ahmed M.Kamel (Other)
Collaborators: The Egyptian IVF-ET Center (Other)
Responsible Party: Sponsor-Investigator, Ahmed M.Kamel, lecturer Of obstetrics & Gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Other Study IDs: 13546
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: anti-Müllerian hormone (AMH); Mullerian anomalies; ICSI
MeSH Terms: conditions — Infertility | interventions — Anti-Mullerian Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mullerian duct anomalies: Anti Mullerian hormone level; Mullerian duct anomaly type
  Interventions: Other: Anti Mullerian hormone level; Mullerian duct anomaly type

INTERVENTIONS:
Other: Anti Mullerian hormone level; Mullerian duct anomaly type — Diagnosis of Mullerian duct anomaly type Clinically or by Imaging Anti-Müllerian Hormone levels

SUMMARY:
Anti-Müllerian hormone (AMH), also known as Müllerian inhibiting substance, is a dimeric glycoprotein that belongs to the transforming growth factor-beta family. It is involved in the regression of the Müllerian ducts during male fetal development. In the female, AMH is solely produced by the granulosa cells of preantral and small antral follicles, and regulates ovarian activity and follicular steroidogenesis

DETAILED DESCRIPTION:
Following approval of the internal review board of Egyptian IVF-ET center, a retrospective analysis will be undertaken where a detailed review of the patients files who underwent intracytoplasmic sperm injection (ICSI) trials starting January 2010 till January 2015 will be done.

Patients with diagnosed mullerian anomalies will have their name , age ,duration of infertility, serum FSH, LH ,& AMH levels recorded. The method of diagnosis (HSG, 3D/ultrasonography, hysteroscopy, or laparoscopy) will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* women with diagnosed mullerian anomlies whether clinically or through imaging

Exclusion Criteria:

* previous ovarian surgery
* ovarian drilling
* polycystic ovarian syndrome (PCOs).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female undergoing intraCytoplasmic sperm injection for treatment of infertility
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Correlation of serum anti-Müllerian hormone (AMH) level with mullerian anomalies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yahia El-fassial, M.D, Principal Investigator — consultant
Locations (1):
- The Egyptian IVF-ET Center, Cairo, Maadi, Egypt

REFERENCES:
- [Background] Li HW, Ng EH, Wong BP, Anderson RA, Ho PC, Yeung WS. Correlation between three assay systems for anti-Mullerian hormone (AMH) determination. J Assist Reprod Genet. 2012 Dec;29(12):1443-6. doi: 10.1007/s10815-012-9880-1. Epub 2012 Nov 2. PMID 23117477